CLINICAL TRIAL: NCT01423526
Title: A Dose Block-randomized, Double-blind, Placebo Controlled, Single-dosing, Dose-escalation Clinical Trial to Investigate the Safety, Tolerability and Pharmacokinetic Characteristics of DWP10292 After Oral Administration in Healthy Male Subjects
Brief Title: A Single Dose Study of DWP10292 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: DWP10292
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2011-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Drug: Placebo tablets, oral administration, single administrations
  Arms: Placebo
  Interventions: Drug: Placebo
- DWP10292 (Experimental): Drug: DWP10292 tablets, oral administration, single administrations
  Arms: DWP10292
  Interventions: Drug: DWP10292

INTERVENTIONS:
Drug: DWP10292 — Drug: DWP10292 tablets, oral administration, single administration
  Arms: DWP10292
Drug: Placebo — Placebo tablets, oral administration, single administrations
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, pharmacokinetics and pharmacodynamics of orally administrated DWP10292 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* A subject who provided written informed consent to participate in this study and cooperative with regard to compliance with study related constraints
* Healthy adult male subjects aged 20 to 45 years
* The subject has a Body weight ≥ 60 kg and < 90 kg and Body Mass Index (BMI) ≥ 18.5 kg/m2 and < 27.0 kg/m2
* A Subject who was judged to be healthy by the investigator to participate in this study based on screening results (according to standard reference index updated recently)

Exclusion Criteria:

* A subject with sign or symptoms or previously diagnosed disease of liver (viral hepatitis), digestive system, cardiovascular, kidney, respiratory, endocrinology, neurology, immune system, hematology, and psychology function or other significant diseases and history or suspicion of current drug abuse and alcohol abuse
* A subject who shows vital signs with the number of systolic blood pressure of ≥140 mmHg or ≤100 mmHg, and the number of diastolic blood pressure of ≥90mmHg or ≤60mmHg
* A subject who shows the following result in clinical laboratory test:

  * AST,ALT>1.25 times of the upper limit of normal range
  * QTc>430msec
  * T.bil>1.25 times of the upper limit of normal range
* A subject from whom over 400mL of blood was sampled(whole blood or plasma donation, etc.) within last 8 weeks
* Subject who has taken other clinical or licensed medication from another clinical trial within an 8-week period prior to the first administration of the study medication (The last administration of the medication is considered as an end point of the previous clinical trial).
* Subject who smokes an average of 10 cigarettes/day and is unable to quit smoking during the clinical trial.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Composite of Pharmacokinetics | 0 (predose), 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 14, 16, 24 (2d 0h), 36, 48 (3d 0h), 60, 72 (4d 0h), 96 h(5d 0h) and Post study visit 216h (10d 0h)
  Cmax, AUClast, AUCinf, Tmax, t1/2, CL/F

SECONDARY OUTCOMES:
Safety&tolerability | 0 (predose), 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 14, 16, 24 (2d 0h), 36, 48 (3d 0h), 60, 72 (4d 0h), 96 h(5d 0h) Post study visit 216h (10d 0h)
  Adverse events, Physical exam, Vital sign, laboratory(CBC,chemistry,U/A etc)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul, Korea
  - Seoul National University Hospital, Seoul